CLINICAL TRIAL: NCT04697979
Title: Post-Stroke Medication Relay
Acronym: REMEDIPA
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL20_0713
Record Dates: First submitted 2021-01-04; First posted 2021-01-06 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2021-01

CONDITIONS: Stroke, Ischemic; Medication Compliance
MeSH Terms: conditions — Ischemic Stroke; Medication Adherence | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire — Selection of patients for a discharge interview in the stroke unit with collection of non-opposition and scheduling of telephone interviews or by teleconsultations at one week and then at two months after hospitalization.
  Data collection through interviews using a telephone questionnaire (or by teleconsultation) one week and then at two months after discharge. Elements on knowledge of treatment, dietary measures and warning signs and recurrence of stroke will be collected and re-explained if necessary.

SUMMARY:
Prior to discharge from hospital and return home, patients managed for ischemic stroke will receive a pharmaceutical interview to discuss their discharge prescription (indication, method of administration, precautions, and possible side effects).

Improvements in the use of medications in the community and in hospital follow-up.

Telephone interviews or teleconsultations will make it possible to assess the patient's knowledge of his or her treatment and to re-explain it if necessary to improve patient compliance with treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients managed in stroke unit following ischemic stroke
* Benefiting from a direct return home
* Non-opposition to participation

Exclusion Criteria:

- None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults patients managed in stroke unit following ischemic stroke who benefiting from a direct return at home.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-02 (Estimated); Primary Completion 2022-02 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Assess the value of a telephone interview / teleconsultation after discharge from hospital following an ischemic stroke | 1 week
  The value of a telephone interview / teleconsultation will be assess by comparison of treatment knowledge between the first questionnaire at one week and the second questionnaire at two months after the pharmaceutical interview and hospital discharge.
  Statistical evaluation by comparative tests at one week versus two months.
  Assessment will focus on treatment knowledge (score between 0 and 3), adherence (score between 0 and 6) and adverse events (score between 0 and 3)
Assess the value of a telephone interview / teleconsultation after discharge from hospital following an ischemic stroke | 2 months
  The value of a telephone interview / teleconsultation will be assess by comparison of treatment knowledge between the first questionnaire at one week and the second questionnaire at two months after the pharmaceutical interview and hospital discharge.
  Statistical evaluation by comparative tests at one week versus two months.
  Assessment will focus on treatment knowledge (score between 0 and 3), adherence (score between 0 and 6) and adverse events (score between 0 and 3)

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Neurologie Vasculaire, Unité 201 Hôpital Neurologique Pierre Wertheimer, HCL, Bron, France

IPD SHARING:
Plan to Share IPD: No